CLINICAL TRIAL: NCT05603780
Title: Cognitive, Emotional, Physiological, Chronobiological and Genetic Effects of a Time Underground Isolation
Brief Title: DEEPTIME: Human Adaptation in Time Underground Isolation
Acronym: DEEPTIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-A00747-37; 27/21_2 (Other: Ethical Committee)
Record Dates: First submitted 2021-12-01; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-08

CONDITIONS: Physiological Stress; Cognitive Dysfunction; Sleep
Keywords: Cognition; exploration; mission; endogenous biological clock; circadian rhythm; adaptation; temporal isolation; free-running; group influence; sleep; temporal anomie
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Follow-up of one group of healthy participant to 40days in a contraint underground environment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group 1 (Other): one cohort
  Interventions: Behavioral: exploratory protocol

INTERVENTIONS:
Behavioral: exploratory protocol — physiological and cognitive evaluations

SUMMARY:
The objectives of this scientific expedition are: a/ Evaluation of temporal cognitive perception and collective synchronization in a temporally anomalous universe (underground environment), b/ Influence of group living on the endogenous circadian rhythmicity of the central biological clock and peripheral clocks in a "free-running" situation (absence of light/natural darkness), c/Evaluation of cognitive and physiological performance in response to exposure to an extreme environment in a natural underground cavity (cave) without access to a time indicator for 40 days, d/Correlation of cognitive, behavioral, psychological, social, neurophysiological and physiological parameters, e/ Determination of adaptation or maladaptation criteria (biological, genetic, physiological, neurophysiological, psychological and cognitive) in an isolation environment (underground) f/ Study of the evolution of collective organization, decision making and leadership in an extreme isolation and management situation.

DETAILED DESCRIPTION:
This exceptional period has shown a significant desynchronization and loss of notion of time in a large number of people as well as important questions about human abilities to live in confined conditions. It is partly for this reason, but also to answer more fundamental questions on the perception of time that the extraordinary research expedition Deep Time was conceived: 40 days underground to know the links of our brain to time and synchronization within a group. A fundamental need for our future. This scientific expedition will take place entirely in France to ensure the feasibility and safety of the subjects and experimenters, under the direction of Christian Clot and the Institute of Human Adaptation, placed under the high patronage of the Ministry of Education, Research and Innovation.

The project addresses the fundamental question of human adaptation to the physical environment and the crucial role of the brain's neuroplasticity properties.

The present "Deep-Time" protocol naturally echoes the "out-of-time" isolation experiments conducted by the speleologist Michel Siffre starting in 1962 and its various components in the years that followed.

These "out of time" experiments led to certain conclusions. As curious as it may seem, in the absence of the time givers (synchronizers or Zeitgebers in German) that are the social rhythms and the day-night alternations, the spontaneous rhythm would settle on a rhythm of about 25 hours.

However, these experiments remained limited to isolated individuals, in conditions of spatial unity (no displacement outside of the work camps), leaving a whole field of research and questioning that the year 2021 has strongly emphasized.

The objectives of this scientific expedition are: a/ Evaluation of temporal cognitive perception and collective synchronization in a temporally anomalous universe (underground environment), b/ Influence of group living on the endogenous circadian rhythmicity of the central biological clock and peripheral clocks in a "free-running" situation (absence of light/natural darkness), c/Evaluation of cognitive and physiological performance in response to exposure to an extreme environment in a natural underground cavity (cave) without access to a time indicator for 40 days, d/Correlation of cognitive, behavioral, psychological, social, neurophysiological and physiological parameters, e/ Determination of adaptation or maladaptation criteria (biological, genetic, physiological, neurophysiological, psychological and cognitive) in an isolation environment (underground) f/ Study of the evolution of collective organization, decision making and leadership in an extreme isolation and management situation.

ELIGIBILITY:
Inclusion Criteria:

Strictly right-handed Good health without any medical and psychiatric diseases No contraindications to MRI French or European nationality Not to be included in another biomedical protocol

Exclusion Criteria:

Being pregnant Minor, under guardianship or curatorship

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-09-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Time | every ten days up to 40 days
  - Evaluation of time perception perceived by subjects (minute and days) every 10 days up to 40 days
chronobiology | every 5 days up to 40 days
  -Influence of group living on the endogenous circadian rhythmicity of the central biological clock and peripheral clocks in a "free-running" situation (absence of light / natural darkness): measurments of body core temperature, cortisol and melatonine salivary concentration circadian rythms
Human Factors: ethological measurments with video 24/24, actimetric circadian rythms | all along the cavern experiment for 40 days
  - Evaluation of the capacity of a group to find a synchronicity and a way of life in a new context, extreme in its environmental and temporal dimensions and out of the initial competences of each group member. Measurments of social interaction, comparison of actimetric circadien rythm
Physiology | every ten days up to 40 days
  Physiological parameters (HRV, lean and fat mass by impedancemtry, weight in kg, core body temperature) in response to exposure to an extreme environment in a natural underground cave for 40 days.
Cognition, Emotion and personnality | every ten to 15 days up to 40 days
  Evaluation of cognitive (taking decision, emotion, spatial cognition) through differents paradigms displayed on screen of Headset in 2D and 3D virtual reality.
  Mesurements of time reaction, risk score, number of strategy or procedural errors, time to achieve the tasks.
  Questionnaires (STAI, POMS, big five inventory, IP9)

CONTACTS AND LOCATIONS:
Overall Officials: stephane besnard, MD, Principal Investigator — CaenHU
Locations (1):
- CHU CAEN, Caen, France

REFERENCES:
- See also: website of the scientific expedition — http://www.deeptime.fr